CLINICAL TRIAL: NCT05719597
Title: Effects of Positive Expiratory Pressure Breathing Versus Incentive Spirometry on Dyspnea and Sputum Profile in Bronchiolectasis Patients
Brief Title: PEP Breathing Versus Incentive Spirometry on Dyspnea and Sputum Profile in Bronchiolectasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0352
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Bronchiolectasis
Keywords: Bronchiolectasis; Dyspnea Severity Index; Incentive Spirometry; Positive Expiratory Pressure (PEP); Saccular Dilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP (Positive Expiratory Pressure) (Experimental): Group A
  Interventions: Other: PEP (Positive Expiratory Pressure)
- IS (Incentive Spirometry) (Experimental): Group B
  Interventions: Other: IS (Incentive spirometry)

INTERVENTIONS:
Other: PEP (Positive Expiratory Pressure) — Group A containing 12 participants, will perform Positive expiratory pressure (PEP) technique for total 60 repetitions (15 repetitions 2 sets, twice) per a day (5 sessions/week and total 4 weeks).
  Arms: PEP (Positive Expiratory Pressure)
Other: IS (Incentive spirometry) — Group B containing 12 participants, will perform Incentive spirometry technique for total 60 repetitions (15 repetitions 2 sets, twice) per a day (5 sessions/week and total 4 weeks).
  Arms: IS (Incentive Spirometry)

SUMMARY:
Bronchiolectasis is the manifestation of chronic bronchitis characterized by saccular dilatation of the terminal bronchioles & bronchiectasis refers to abnormal dilatation of the bronchi. In bronchiolectasis more proximal bronchi may or may not show radiological changes. Airway dilatation can lead to failure of mucus clearance and increased risk of infection. Pathophysiological mechanism of bronchiectasis/bronchiolectasis include persistent bacterial infections, deregulated immune responses, impaired mucociliary clearance and airway obstruction. Treatment is directed at reducing the frequency of exacerbations, improving quality of life. Although no therapy is licensed for bronchiectasis by regulatory agencies, evidence supports the effectiveness of airway clearance techniques, antibiotics and mucolytic agents. Enhancing effective expectoration of stagnated bronchopulmonary secretions, usually with physiotherapy support, is key to management. There are different methods for delivering chest physiotherapy, such as the active cycle of breathing technique, postural drainage, (PEP) and oscillating PEP devices. The objective of the study is to compare the effects of PEP & Incentive spirometry techniques on bronchiolectasis patients.

The study will be a randomized clinical trial. Total 24 subjects will be assigned randomly into two groups by using convenient sampling technique. Baseline treatment will be same (chest physiotherapy) in both groups. Group A will use PEP and Group B will use incentive spirometry technique for total 60 repetitions (15 repetitions 2 sets, two times per a day) 5 sessions per week and total 4 weeks. Dyspnea severity index and cough & sputum assessment questionnaire (CASA-Q) would be used as an outcome measurement tools. Measurements will be taken at Baseline, and at the end of the 4 weeks treatment session. After assessing the normality, data will be analyzed by using parametric and non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 22 to 85 years
* Both GenderCOVID-19 negative
* Indoor patients
* Ability to use PEP devices
* Diagnosed Bronchiolectasis Patients (through CT scan, X-Ray)

Exclusion Criteria:

* Rib fracture
* Neurological problems
* Lungs carcinomas
* Any other serious comorbidity

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea Severity Index | 4 Weeks
  The Dyspnea severity index is a patient-centered questionnaire that can be used for assessment of initial severity of dyspnea symptoms related to the upper airway and can also be used as a follow-up assessment tool to evaluate treatment outcomes and drive evidence-based medical decisions.
Cough and Sputum Assessment Questionnaire (CASA-Q) | 4 Weeks
  The CASA-Q is a self-administered questionnaire that assesses cough and sputum based on their frequency, severity, and impact on daily activities in the previous 7 days. The CASA-Q contains four domains: cough symptoms, cough impact, sputum symptoms, and sputum impact.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson WH, Coakley RD, Button B, Henderson AG, Zeman KL, Alexis NE, Peden DB, Lazarowski ER, Davis CW, Bailey S, Fuller F, Almond M, Qaqish B, Bordonali E, Rubinstein M, Bennett WD, Kesimer M, Boucher RC. The Relationship of Mucus Concentration (Hydration) to Mucus Osmotic Pressure and Transport in Chronic Bronchitis. Am J Respir Crit Care Med. 2015 Jul 15;192(2):182-90. doi: 10.1164/rccm.201412-2230OC. PMID 25909230
- [Background] King PT. The pathophysiology of bronchiectasis. Int J Chron Obstruct Pulmon Dis. 2009;4:411-9. doi: 10.2147/copd.s6133. Epub 2009 Nov 29. PMID 20037680
- [Background] WISOFF CP. Bronchiolectasis in chronic bronchitis. Radiology. 1958 Jun;70(6):848-50. doi: 10.1148/70.6.848. No abstract available. PMID 13554852
- [Background] Redondo M, Keyt H, Dhar R, Chalmers JD. Global impact of bronchiectasis and cystic fibrosis. Breathe (Sheff). 2016 Sep;12(3):222-235. doi: 10.1183/20734735.007516. PMID 28210295
- [Background] King PT, Holdsworth SR, Freezer NJ, Villanueva E, Holmes PW. Characterisation of the onset and presenting clinical features of adult bronchiectasis. Respir Med. 2006 Dec;100(12):2183-9. doi: 10.1016/j.rmed.2006.03.012. Epub 2006 May 2. PMID 16650970
- [Background] Dodd JD, Lavelle LP, Fabre A, Brady D. Imaging in cystic fibrosis and non-cystic fibrosis bronchiectasis. Semin Respir Crit Care Med. 2015 Apr;36(2):194-206. doi: 10.1055/s-0035-1546749. Epub 2015 Mar 31. PMID 25826587
- [Background] Chalmers JD, Chang AB, Chotirmall SH, Dhar R, McShane PJ. Bronchiectasis. Nat Rev Dis Primers. 2018 Nov 15;4(1):45. doi: 10.1038/s41572-018-0042-3. PMID 30442957
- [Background] Lee AL, Williamson HC, Lorensini S, Spencer LM. The effects of oscillating positive expiratory pressure therapy in adults with stable non-cystic fibrosis bronchiectasis: A systematic review. Chron Respir Dis. 2015 Feb;12(1):36-46. doi: 10.1177/1479972314562407. Epub 2014 Dec 17. PMID 25518845
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] Reychler G, Uribe Rodriguez V, Hickmann CE, Tombal B, Laterre PF, Feyaerts A, Roeseler J. Incentive spirometry and positive expiratory pressure improve ventilation and recruitment in postoperative recovery: A randomized crossover study. Physiother Theory Pract. 2019 Mar;35(3):199-205. doi: 10.1080/09593985.2018.1443185. Epub 2018 Feb 27. PMID 29485340